CLINICAL TRIAL: NCT04675788
Title: Novel Approaches for Minimizing Drug-Induced QT Interval Lengthening
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Purdue University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Harvard University (Other); Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, James E. Tisdale, Professor of PharmD, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005890134; 1R01HL153114-01 (NIH)
Record Dates: First submitted 2020-12-04; First posted 2020-12-19 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Long QT Syndrome; Abnormalities, Drug-Induced
MeSH Terms: conditions — Long QT Syndrome; Abnormalities, Drug-Induced | interventions — Progesterone; ibutilide; Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Postmenopausal women: Progesterone (Experimental): Subjects will receive treatment with oral progesterone 400 mg once daily (two x 200 mg capsules) every evening for 7 days
  Interventions: Drug: Progesterone; Drug: Ibutilide
- Postmenopausal women: Placebo (Placebo Comparator): Subjects will receive oral placebo, two capsules once daily every evening for 7 days
  Interventions: Drug: Ibutilide; Drug: Placebo
- Men 65 years of age or older: Testosterone (Experimental): Subjects will receive treatment with transdermal testosterone 1% (100 mg) every morning for 3 days
  Interventions: Drug: Ibutilide; Drug: Testosterone
- Men 65 years of age or older: Placebo (Placebo Comparator): Subjects will receive treatment with transdermal placebo every morning for 3 days
  Interventions: Drug: Ibutilide; Drug: Placebo

INTERVENTIONS:
Drug: Progesterone — Subjects will receive oral progesterone 400 mg (two x 200 mg capsules) once daily every evening for 7 days
  Arms: Postmenopausal women: Progesterone
Drug: Ibutilide — Ibutilide 0.003 mg/kg administered to all subjects to modestly lengthen the QT interval
  Other Names: Corvert
Drug: Testosterone — Subjects will apply transdermal testosterone gel once daily every morning for 3 days
  Other Names: Androgel
  Arms: Men 65 years of age or older: Testosterone
Drug: Placebo — Lactose capsules
  Arms: Men 65 years of age or older: Placebo; Postmenopausal women: Placebo

SUMMARY:
This research will determine if: 1) Oral progesterone attenuates drug-induced QT interval, J-Tpeak and Tpeak-Tend lengthening in postmenopausal women 50 years of age or older, and 2) Transdermal testosterone attenuates drug-induced QT interval, J-Tpeak and Tpeak-Tend lengthening in men 65 years of age or older. This investigation will consist of two concurrent prospective, randomized, double-blind, placebo-controlled crossover-design studies in a) Postmenopausal women, and b) Men 65 years of age or older. Study 1: Each postmenopausal woman will take progesterone or placebo capsules for 1 week. After a 14-day "washout" (no progesterone or placebo) each subject will then take the alternative therapy (progesterone or placebo) for 1 week. After 7 days of each treatment, subjects will present to the clinical research center to receive a small dose of the QT interval-lengthening drug ibutilide, and the effect on the QT, J-Tpeak and Tpeak-Tend intervals during the progesterone and placebo phases will be compared. Study 2: Each man 65 years of age or older will apply transdermal testosterone or transdermal placebo gel for 3 days. After a 7-day "washout" (no testosterone or placebo) each subject will then apply the alternative therapy (testosterone or placebo gel) for 1 week. After 3 days of each treatment, subjects will present to the clinical research center to receive a small dose of the QT interval-lengthening drug ibutilide, and the effect on the QT, J-Tpeak and Tpeak-Tend intervals during the testosterone and placebo phases will be compared.

DETAILED DESCRIPTION:
Torsades de pointes (TdP) is a ventricular tachycardia associated with prolongation of the corrected QT (QTc) interval, and which may be caused by > 150 widely used drugs. TdP results in catastrophic outcomes, including sudden cardiac death. Older age is a risk factor for drug-induced TdP, possibly due to declining serum progesterone and testosterone concentrations in postmenopausal women and men, respectively. The ECG biomarkers J-Tpeak and Tpeak-Tend, represent early and late repolarization, respectively, as well as dispersion of repolarization (Tpeak-Tend). Preclinical evidence and preliminary data from our group indicate that progesterone and testosterone exert protective effects against drug-induced prolongation of ventricular repolarization. Effective means of reducing the risk of drug-induced QTc interval prolongation and TdP in high risk populations requiring therapy with QTc-prolonging drugs have not been identified, and the effects of sex hormones on early vs late ventricular repolarization and dispersion of repolarization are unknown. The objectives of this research are to evaluate novel therapeutic approaches to attenuate drug-induced QTc lengthening. Our central hypothesis is that drug-induced QTc lengthening is attenuated by administration of oral progesterone and transdermal testosterone. Specific Aim 1: Determine the efficacy of oral progesterone as a preventive method to attenuate drug-induced QTc interval lengthening in postmenopausal women. Specific Aim 2: Determine the efficacy of transdermal testosterone as a preventive method to attenuate drug-induced QTc interval lengthening in men ≥ 65 years of age. Specific Aim 3a: Determine the influence of oral progesterone on drug-induced lengthening of early and late ventricular repolarization in postmenopausal women. Specific Aim 3b: Determine the influence of transdermal testosterone on drug-induced lengthening of early and late ventricular repolarization in men ≥ 65 years of age. Specific Aims 1&3a will be achieved via a prospective, randomized, double-blind, placebo-controlled two-way crossover study in postmenopausal women age ≥ 50 years (n=48). Each subject will take oral progesterone 400 mg or matching placebo daily for 7 days (≥ 14-day washout period between phases). On day 7, each subject will receive a single dose of the QTc-lengthening drug ibutilide 0.003 mg/kg. Specific Aims 2&3b will be achieved via a prospective, randomized, double-blind, placebo-controlled two-way crossover study in men ≥ 65 years of age (n=35). Each subject will apply transdermal testosterone 1% 100 mg or transdermal placebo once daily for 3 days (≥ 7-day washout period between phases). On day 7, each subject will ibutilide 0.003 mg/kg. In both studies, post-ibutilide QT, J-Tpeak and Tpeak-Tend intervals and serum ibutilide concentrations will be determined serially. Primary outcome measures: 1) Maximum post-ibutilide QTc intervals, 2) Maximum post-ibutilide % change in QTc intervals, 3) Area under the QTc interval-time curves, and 4) J-Tpeak and Tpeak-Tend intervals. This research will identify effective approaches for reducing the risk of drug-induced QTc interval prolongation in high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal Women:

* Age 50-99 years old
* Postmenopausal (have not has a menstrual period for 12 months or longer)

Exclusion Criteria:

Postmenopausal women:

* Subject reported history of breast, uterine and ovarian cervical cancer
* Subject reported history of hysterectomy and/or ovariectomy
* Subject reported taking any hormone replacement therapy (prescription, nonprescription or herbal supplement)
* Weight < 60 kg at time of screening visit
* Weight >135 kg at time of screening visit
* Serum K+ <3.6 mEq/L at time of any ibutilide dosing visit
* Serum Mg2+ <1.8 mg/dL at time of screening visit
* Hematocrit <26%
* AST or ALT > 3x the upper limit of normal (determined by testing lab ranges) at the time of screening visit
* Baseline Bazett's-corrected QTc >450 ms (during any visit prior to ibutilide dosing)
* Baseline QRS > 120 ms (at time of baseline visit)
* Diagnosis of heart failure due to reduced or preserved ejection fraction
* Subject reported family history of long QT syndrome, TdP, or sudden cardiac death not associated with acute myocardial infarction
* Self-reported personal history of long QT syndrome, sudden cardiac death not associated with acute myocardial infarction
* Subject reported history any prolonged arrhythmia for which treatment was required
* Subject reported history of a myocardial infarction
* Subject reported history of coronary artery disease
* Sustained arrythmia found at baseline screening prior to any study visit including atrial fibrillation, atrial flutter, junctional rhythm, heart block (any)
* Permanently paced ventricular rhythm
* Current reported use of any QT prolonging medication. Investigator will check the current QT drugs list at www.crediblemeds.org during screening.
* Current reported use of any moderate or strong inhibitors of cytochrome P450 (CYP) 3A4, 3A5, or 3A7
* Current reported use of any inducers of cytochrome P-450 (CYP) 3A4, 3A5 or 3A7

Inclusion Criteria:

Older Men:

• Age 65 years old to 99 years old

Exclusion Criteria:

* Older men:
* Subject reported diagnosis of benign prostatic hyperplasia
* Subject reported history of breast or prostate cancer
* Weight < 60 kg at time of screening visit
* Weight >135 kg at time of screening visit
* Serum K+ <3.6 mEq/L at time of any ibutilide dosing visit
* Serum Mg2+ <1.8 mg/dL at time of screening visit
* Hematocrit <26%
* AST or ALT > 3x the upper limit of normal (determined by testing lab ranges) at the time of screening visit
* Baseline Bazett's-corrected QTc >450 ms (during any visit prior to ibutilide dosing)
* Baseline QRS > 120 ms (at time of baseline visit)
* Diagnosis of heart failure due to reduced or preserved ejection fraction
* Subject reported family history of long QT syndrome, TdP, or sudden cardiac death not associated with acute myocardial infarction
* Self-reported personal history of long QT syndrome, arrhythmias (including atrial fibrillation) or sudden cardiac death not associated with acute myocardial infarction
* Sustained arrythmia found at baseline screening prior to any study visit including atrial fibrillation, atrial flutter, junctional rhythm, heart block (any)
* Permanently paced ventricular rhythm
* Current reported use of any QT prolonging medication (Investigator will check current list of QT prolonging medications listed at www.crediblemeds.org at the time of screening for the most up to date list.
* Current reported use of any moderate or strong inhibitors of cytochrome P450 (CYP) 3A
* Current reported use of any inducers of cytochrome P-450 (CYP) 3A4, 3A5 or 3A7

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Pre-ibutilide QT-F and QT-Fram intervals | Morning of day 8 (after 7 days of progesterone/placebo)
  QT intervals will be corrected for heart rate using two methods: the Fridericia method and the Framingham method
Pre-ibutilide QT-F and QT-Fram intervals | Morning of day 4 (after 3 days of testosterone/placebo)
  QT intervals will be corrected for heart rate using two methods: the Fridericia method and the Framingham method
Maximum post-ibutilide QT-F and QT-Fram intervals | From initiation of ibutilide infusion and for 8 hours after the end of ibutilide infusion
  Maximum post-ibutilide QT-F and QT-Fram intervals
Percent change from baseline (pre-ibutilide) in maximum QT-F and QT-Fram intervals | From initiation of ibutilide infusion and for 8 hours after the end of ibutilide infusion
  Percent change from baseline (pre-ibutilide) in maximum QT-F and QT-Fram intervals
Area under the QT-F and QT-Fram versus time curves during and for 1 hour following ibutilide infusion | From initiation of ibutilide infusion and for 1 hour after the end of ibutilide infusion
  Area under the QT-F and QT-Fram versus time curves during and for 1 hour
Area under the QT-F and QT-Fram versus time curves during and for 8 hours following ibutilide infusion | From initiation of ibutilide infusion and for 8 hours after the end of ibutilide infusion
  Area under the QT-F and QT-Fram versus time curves during and for 8 hours following ibutilide infusion
Pre-ibutilide heart rate-corrected J-Tpeak (J-Tpeakc) intervals | Morning of day 8 (after 7 days of progesterone/placebo)
  Pre-ibutilide heart rate-corrected J-Tpeak (J-Tpeakc) intervals
Pre-ibutilide heart rate-corrected J-Tpeak (J-Tpeakc) intervals | Morning of day 4 (after 3 days of testosterone/placebo)
  Pre-ibutilide heart rate-corrected J-Tpeak (J-Tpeakc) intervals
Maximum post-ibutilide J-Tpeakc intervals | From initiation of ibutilide infusion and for 8 hours after the end of ibutilide infusion
  Maximum post-ibutilide J-Tpeakc intervals
Percent change from baseline (pre-ibutilide) in maximum J-Tpeakc intervals | From initiation of ibutilide infusion and for 8 hours after the end of ibutilide infusion
  Percent change from baseline (pre-ibutilide) in maximum J-Tpeakc intervals
Area under the J-Tpeakc versus time curve during and for 1 hour following ibutilide infusion | From initiation of ibutilide infusion and for 1 hour after the end of ibutilide infusion
  Area under the J-Tpeakc versus time curve during and for 1 hour following ibutilide infusion
Area under the J-Tpeakc versus time curve during and for 8 hours following ibutilide infusion | From initiation of ibutilide infusion and for 8 hours after the end of ibutilide infusion
  Area under the J-Tpeakc versus time curve during and for 8 hours following ibutilide infusion
Pre-ibutilide Tpeak-Tend intervals | Morning of day 8 (after 7 days of progesterone/placebo)
  Pre-ibutilide Tpeak-Tend intervals
Pre-ibutilide Tpeak-Tend intervals | Morning of day 4 (after 3 days of testosterone/placebo)
  Pre-ibutilide Tpeak-Tend intervals
Maximum post-ibutilide Tpeak-Tend intervals | From initiation of ibutilide infusion and for 8 hours after the end of ibutilide infusion
  Maximum post-ibutilide Tpeak-Tend intervals
Percent change from baseline (pre-ibutilide) maximum Tpeak-Tend intervals | From initiation of ibutilide infusion and for 8 hours after the end of ibutilide infusion
  Percent change from baseline (pre-ibutilide) maximum Tpeak-Tend intervals
Area under the Tpeak-Tend versus time curves during and for 1 hour following ibutilide infusion | From initiation of ibutilide infusion and for 1 hour after the end of ibutilide infusion
  Area under the Tpeak-Tend versus time curves during and for 1 hour following ibutilide infusion
Area under the Tpeak-Tend versus time curves during and for 8 hours following ibutilide infusion | From initiation of ibutilide infusion and for 8 hours after the end of ibutilide infusion
  Area under the Tpeak-Tend versus time curves during and for 8 hours following ibutilide infusion

OTHER OUTCOMES:
Adverse effects of oral progesterone and placebo | Adverse effects will be assessed via telephone calls to subjects between days 2 and 4 and between days 5 and 7 of oral progesterone and oral placebo
  Adverse effects of oral progesterone and oral placebo
Adverse effects of transdermal testosterone and transdermal placebo | Adverse effects will be assessed via telephone calls to subjects between days 1 and 3 of transdermal testosterone and transdermal placebo
  Adverse effects of transdermal testosterone and transdermal placebo
Adverse effects of ibutilide | Adverse effects of ibutilide will be assessed during the 10-minute intravenous infusion and for 8 hours following the infusion of ibutilide
  Adverse effects of ibutilide

CONTACTS AND LOCATIONS:
Overall Officials: James E Tisdale, PharmD, Principal Investigator — Purdue University
Locations (3):
- United States (3):
  - Indiana Clinical Research Center, Indianapolis, Indiana
  - Indiana University, Indianapolis, Indiana
  - Purdue University, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No